CLINICAL TRIAL: NCT06202872
Title: Memory Enhancement Using Transcranial Alternating Current Stimulation
Acronym: Memento
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Willem de Haan, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20212222
Record Dates: First submitted 2023-12-22; First posted 2024-01-12 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-09

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
Keywords: Alzheimer's disease; Transcranial alternating current stimulation; Episodic memory; Magnetoencephalography
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomized, sham-controlled, crossover trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active tACS (Experimental): Gamma (40 Hz) tACS at the precuneus region
  Interventions: Device: Gamma (40 Hz) tACS at the precuneus region
- Sham tACS (Sham Comparator): Sham tACS at the precuneus region
  Interventions: Device: Sham tACS at the precuneus region

INTERVENTIONS:
Device: Gamma (40 Hz) tACS at the precuneus region — 40 Hz tACS applied at a current of 3.2 milliampere peak-to-peak using a NuroStym transcranial electrical stimulation (tES) system of NeuroDevice for four times 12 minutes (48 minutes in total) at the Pz (according to the 10-20 international EEG coordinates)
  Arms: Active tACS
Device: Sham tACS at the precuneus region — Sham tACS applied with no effective stimulation between the ramp-up and ramp-down of the current using a NuroStym tES system of NeuroDevice for four times 12 minutes (48 minutes in total) at the Pz (according to the 10-20 international EEG coordinates)
  Arms: Sham tACS

SUMMARY:
The 32 million Alzheimer's disease (AD) and 69 million prodromal AD patients worldwide contribute to a large economic burden. Effective and safe therapies that slow or prevent the progression from mild cognitive impairment (MCI) to AD are therefore of high priority. Transcranial alternating current stimulation (tACS) is a safe and patient-friendly non-invasive brain stimulation technique that serves as a potential candidate for reducing and/or slowing cognitive impairment. Application of tACS in the gamma frequency range, specifically around 40 Hz, has been studied in patients with AD and MCI due to AD. In these patients, a single session of 40 Hz tACS at the precuneus showed to improve episodic memory and to increase gamma power, as measured with electroencephalography. These findings will be replicated in the current study in patients with MCI due to AD, using magnetoencephalography (MEG) recorded before, during and after tACS. In this way, brain activity and network changes that underlie this improvement in episodic memory can be studied with greater temporal and spatial detail.

ELIGIBILITY:
Inclusion Criteria:

* Recent (not more than 6 months ago) amnestic MCI diagnosis, which consensus is obtained in a multidisciplinary meeting after an extended multidisciplinary test battery at the memory clinic, including confirmation of AD pathology with cerebrospinal fluid biomarkers: abnormal p-tau/Aβ42 ratio of > 0.023

Exclusion Criteria:

* Suffering from serious neurological, psychiatric or somatic comorbidity
* Suffering from epileptic seizures or severe claustrophobia
* Intensive use of psychoactive medication
* Having a cardiac pacemaker, internal cardiac defibrillator or other intracorporeal device that interferes with MEG recordings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Rey Auditory Verbal Learning test scores | Immediately before and after intervention
  The Rey Auditory Verbal Learning (RAVL) test evaluates verbal episodic memory and is designed as a list-learning paradigm in which the subject hears a list of 15 nouns. The participant is asked to recall as many words from the list as possible after each of 5 repetitions of free-recall (total recall), and 15 minutes after an interference trial (long delayed recall). Scores range from 0 to 75 (total recall) and 0 to 15 (long delayed recall), with higher scores meaning a better outcome. An increase in RAVL test (total and long delayed recall) after active but not sham tACS is expected.
Change in Face-Name Association Task scores | Immediately before and after intervention
  The Face-Name Association Task assesses associative episodic memory and is a computer paradigm consisting of an encoding and a retrieval phase of face-name pairs. During the encoding phase, participants are instructed to remember a set of 12 faces and names they are paired. In two additional learning trials, participants are shown the previously learned faces and are asked to recall the correct name associated with each face (inital recognition). This recall of the correct name associated with a learned face is repeated 5 minutes after the learning trials during the retrieval phase (associative recognition). Scores range from 0 to 24 (inital recognition) and 0 to 12 (associative recognition), with higher scores meaning a better outcome. An increase in FNAT score (initial and associative recognition) after active but not sham tACS is expected.

SECONDARY OUTCOMES:
Change in spectral source space resting-state MEG (relative power) | Immediately before and after intervention
  Change in relative power will be used, expecting an increase in relative power in higher alpha, beta and gamma bands and decrease in relative power in theta band after active but not sham tACS.
Change in spectral source space resting-state MEG (posterior peak frequency) | Immediately before and after intervention
  Change in posterior peak frequency will be used, expecting an increase in posterior peak frequency after active but not sham tACS.
Change in functional connectivity source space resting-state MEG (AEC-c) | Immediately before and after intervention
  Change in corrected amplitude envelope correlation (AEC-c) will be used, expecting an increase in AEC-c in higher alpha, beta and gamma bands after active but not sham tACS.
Change in functional connectivity source space resting-state MEG (PLI) | Immediately before and after intervention
  Change in phase lag index (PLI) will be used, expecting a decrease in PLI in theta band after active but not sham tACS.
Change in source space resting-state MEG network structure (MST variables) | Immediately before and after intervention
  Change in graph theory parameters will be used as a measure of global network structure. Restoration of overall network configuration (expressed by shift of multiple Minimum spanning tree (MST) parameters towards healthy state, e.g. stronger hierarchy) after active but not sham tACS is expected.
Change in source space resting-state MEG network structure (clustering coefficient and path length) | Immediately before and after intervention
  Change in graph theory parameters will be used as a measure of global network structure. Preserved small-world configuration (shift of small world index (clustering coefficient/path length) towards less random topology) after active but not sham tACS is expected.
Change in source space resting-state MEG network structure (modulatory index, degree and eigenvector centrality) | Immediately before and after intervention
  Change in graph theory parameters will be used as a measure of mesoscale network structure (modularory measures) and nodal characteristics (degree and eigenvector centrality). Restoration of hub disruption (stronger modularity index, increase in degree and eigenvector centrality) of precuneus-posterior cingulate and medial temporal lobe after active but not sham tACS is expected.

CONTACTS AND LOCATIONS:
Overall Officials: Willem de Haan, dr., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Amsterdam UMC, The Netherlands, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data will be made available upon reasonable request to the corresponding author in consultation with the data protection officer
Time Frame: Data will be shared after the study completion indefinitely
Access Criteria: Upon reasonable request

REFERENCES:
- [Background] Benussi A, Cantoni V, Cotelli MS, Cotelli M, Brattini C, Datta A, Thomas C, Santarnecchi E, Pascual-Leone A, Borroni B. Exposure to gamma tACS in Alzheimer's disease: A randomized, double-blind, sham-controlled, crossover, pilot study. Brain Stimul. 2021 May-Jun;14(3):531-540. doi: 10.1016/j.brs.2021.03.007. Epub 2021 Mar 21. PMID 33762220
- [Background] Benussi A, Cantoni V, Grassi M, Brechet L, Michel CM, Datta A, Thomas C, Gazzina S, Cotelli MS, Bianchi M, Premi E, Gadola Y, Cotelli M, Pengo M, Perrone F, Scolaro M, Archetti S, Solje E, Padovani A, Pascual-Leone A, Borroni B. Increasing Brain Gamma Activity Improves Episodic Memory and Restores Cholinergic Dysfunction in Alzheimer's Disease. Ann Neurol. 2022 Aug;92(2):322-334. doi: 10.1002/ana.26411. Epub 2022 Jun 6. PMID 35607946
- [Background] Grover S, Fayzullina R, Bullard BM, Levina V, Reinhart RMG. A meta-analysis suggests that tACS improves cognition in healthy, aging, and psychiatric populations. Sci Transl Med. 2023 May 24;15(697):eabo2044. doi: 10.1126/scitranslmed.abo2044. Epub 2023 May 24. PMID 37224229
- [Background] Iaccarino HF, Singer AC, Martorell AJ, Rudenko A, Gao F, Gillingham TZ, Mathys H, Seo J, Kritskiy O, Abdurrob F, Adaikkan C, Canter RG, Rueda R, Brown EN, Boyden ES, Tsai LH. Gamma frequency entrainment attenuates amyloid load and modifies microglia. Nature. 2016 Dec 7;540(7632):230-235. doi: 10.1038/nature20587. PMID 27929004
- [Background] Maestu F, de Haan W, Busche MA, DeFelipe J. Neuronal excitation/inhibition imbalance: core element of a translational perspective on Alzheimer pathophysiology. Ageing Res Rev. 2021 Aug;69:101372. doi: 10.1016/j.arr.2021.101372. Epub 2021 May 21. PMID 34029743
- [Background] Palop JJ, Mucke L. Network abnormalities and interneuron dysfunction in Alzheimer disease. Nat Rev Neurosci. 2016 Dec;17(12):777-792. doi: 10.1038/nrn.2016.141. Epub 2016 Nov 10. PMID 27829687